CLINICAL TRIAL: NCT01237743
Title: Transcranial Doppler Microembolic Signals and Serum Markers of Neuronal Damage During Transcatheter Aortic Valve Implantation
Brief Title: Microembolic Signals and Serum Markers of Neuronal Damage During Transcatheter Aortic Valve Implantation.
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Professor Sven Erik Ricksten, Sahlgrenska University Hospital. The sahlgrenska Academy.Institution Of Thoracic Anaesthesia & Intensive Care,Gothenburg Sweden
Other Study IDs: Dnr304-09
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2010-11

CONDITIONS: Aortic Stenosis
Keywords: Embolism; Nervous system; Aorta; Valves; Ultrasonics
MeSH Terms: conditions — Aortic Valve Stenosis; Embolism; Neurologic Manifestations | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum levels of S-100β Determined by an electrochemoluminescence immunoassay using the Modular system and the S100β reagent kit (Roche Diagnostics, Basel, Switzerland).
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Transcatheter aortic valve implantation. — Transcatheter aortic valve implantation,femoral access.
  Other Names: Core Valve ® (Medtronic, Inc., Minneapolis, Minnesota)

SUMMARY:
Transcatheter Aortic Valve Implantation (TAVI) using femoral access is an option for definitive treatment of aortic stenosis when open-heart surgery is considered inappropriate. By avoiding the effects of cardiopulmonary bypass on cerebral hemodynamics and microembolic load, TAVI is assumed to be beneficial regarding risk for neurological complications. We anticipated that the extensive endovascular retrograde manipulation in ascending aorta and aortic root would generate a detectable cerebral microembolic load, and thus an increase in serological markers of neuronal injury postoperatively. Our hypothesis is that there is a positive correlation between the total amount of cerebral microembolic events during the TAVI procedure and the Area under curve (AUC24hrs) for the release pattern of two markers of neuronal injury. We also wish to describe the extent and distribution of microembolisms during the TAVI procedure using Transcranial Doppler (TCD).

DETAILED DESCRIPTION:
Patients scheduled for TAVI at our institution are screened for inclusion into this prospective, observational study. A multidisciplinary expert committee evaluate all high-risk patients diagnosed with aortic stenosis. If rejected for open-heart surgery, and without contraindications for transcatheter approach, the patient is offered treatment with TAVI using the CoreValve ® (Medtronic, Inc., Minneapolis, Minnesota) system. The Human Ethics Committee of the University of Gothenburg, approved the study protocol, and all patients sign an informed, written consent. CoreValve ® is a TAVI system delivering a tri-leaflet bioprosthetic porcine pericardial tissue valve mounted and sutured in a self-expanding nitinol frame, using a trans-femoral or trans-subclavian artery access approach. Details regarding the TAVI procedure have been described previously . On the evening before surgery, the patients receive a loading dose of clopidogrel 300 mg. The morning of surgery an additional dose of clopidogrel 75 mg, together with acetylsalicylic acid 75 mg is given.

No sedative premedication is given before the procedure. On arrival at OR, standard perioperative monitoring is established, including an Auditory Evoked Potential (AEP) monitor for anaesthetic depth measurements (AEP Monitor/2, Danmeter, Odense, Denmark) and radial arterial and central venous lines. General anaesthesia is induced with propofol 0.5-1 mg/kg and fentanyl 100-150 μg. Tracheal intubation facilitated using atracurium 0,5 mg/kg. A propofol infusion is used to maintain an anaesthetic depth adjusted to an AAI index of 15-30 as recorded by the AEP monitor. Hemodynamic stability is obtained by the use of colloidal solution administration, guided by the use of intra-operative transesophageal echocardiography, and norephineprine to maintain a mean arterial pressure above 75 mmHg. During the procedure, intravenous heparin is administered to achieve an activated clotting time > 250 sec. Catheters and guide-wires are flushed and cleaned according to standard procedures at our laboratory. The preparation of the valve is performed according to the instructions of the manufacturer. The balloon valvuloplasty of the native aortic valve is performed under rapid right ventricular pacing (180 bpm) and the self-expandable prosthesis deployed stepwise without pacing. The same team of two interventional cardiologists and one cardiothoracic anaesthesiologist perform all procedures. A certified cardiologist or anaesthesiologist assess focal neurological impairment before and within 24 hours after the procedure.

ELIGIBILITY:
Inclusion Criteria: Clinical diagnosis of Aortic stenosis rejected for open-heart surgery.

-

Exclusion Criteria: None

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with aortic stenosis rejected for open-heart surgery due to unacceptable risks.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Transcranial Doppler microembolic signals during transcatheter aortic valve implantation | During surgery

SECONDARY OUTCOMES:
Area under curve for the release pattern of serum S-100β after transcatheter aortic valve implantation | 24 Hour after Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sven Erik Ricksten, Professor, Study Director — Sahlgrenska University Hospital,Thoracic Anesthesia & Intensive Care
Locations (1):
- Department of Thoracic Anaesthesia & Intensive Care,Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Dittrich R, Ringelstein EB. Occurrence and clinical impact of microembolic signals during or after cardiosurgical procedures. Stroke. 2008 Feb;39(2):503-11. doi: 10.1161/STROKEAHA.107.491241. Epub 2008 Jan 3. PMID 18174490
- [Background] Lund C, Nes RB, Ugelstad TP, Due-Tonnessen P, Andersen R, Hol PK, Brucher R, Russell D. Cerebral emboli during left heart catheterization may cause acute brain injury. Eur Heart J. 2005 Jul;26(13):1269-75. doi: 10.1093/eurheartj/ehi148. Epub 2005 Feb 16. PMID 15716287
- [Background] Webb JG, Pasupati S, Humphries K, Thompson C, Altwegg L, Moss R, Sinhal A, Carere RG, Munt B, Ricci D, Ye J, Cheung A, Lichtenstein SV. Percutaneous transarterial aortic valve replacement in selected high-risk patients with aortic stenosis. Circulation. 2007 Aug 14;116(7):755-63. doi: 10.1161/CIRCULATIONAHA.107.698258. Epub 2007 Jul 23. PMID 17646579
- [Derived] Reinsfelt B, Westerlind A, Ioanes D, Zetterberg H, Freden-Lindqvist J, Ricksten SE. Transcranial Doppler microembolic signals and serum marker evidence of brain injury during transcatheter aortic valve implantation. Acta Anaesthesiol Scand. 2012 Feb;56(2):240-7. doi: 10.1111/j.1399-6576.2011.02563.x. Epub 2011 Oct 19. PMID 22092012